CLINICAL TRIAL: NCT00134875
Title: Abuse Potential of Parenteral Buprenorphine/Naloxone in Non-Dependent Opioid Abusers
Brief Title: Assessing Abuse Potential of Parenteral Buprenorphine/Naloxone in Non-Dependent Opioid Abusers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Eric C. Strain/Principal Investigator, Johns Hopkins University School of Medicine
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08045-3; R01-08045-3; DPMC
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-10

CONDITIONS: Opioid-Related Disorders
Keywords: opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Acute doses of buprenorphine/naloxone in each experimental test session. Doses delivered by either sublingual or parenteral routes, and are: 4/1, 8/2, 16/4 mg.

SUMMARY:
Buprenorphine, a treatment for opioid dependence, can be mixed with another drug, naloxone, to limit abuse potential. Parenteral administration (intravenous or intramuscular injection) of buprenorphine/naloxone causes withdrawal symptoms in opioid dependent individuals. However, naloxone does not cause withdrawal symptoms in non-dependent opioid abusers. This study will investigate whether naloxone decreases the opioid agonist effect from injected buprenorphine, hence decreasing the abuse potential of buprenorphine/naloxone, in non-dependent opioid abusers.

DETAILED DESCRIPTION:
Naloxone has been combined with buprenorphine to decrease the parenteral abuse potential of buprenorphine in opioid dependent individuals through the mechanism of naloxone-precipitated withdrawal. While naloxone will not precipitate withdrawal in individuals who are not physically dependent on opioids, it is possible naloxone might attenuate buprenorphine's agonist effects, especially if administered parenterally. The purpose of this study is to assess the effect of sublingual (SL) and intramuscular (IM) buprenorphine and buprenorphine/naloxone in non-dependent opioid abusers.

Participants will stay on a research ward and will undergo challenge sessions twice per week. The following conditions will be tested: placebo; IM hydromorphone (2 and 4 mg; an opioid agonist positive control condition); SL buprenorphine (4, 8, and 16 mg); IM buprenorphine (4, 8, and 16 mg); SL buprenorphine/naloxone(4/1, 8/2, and 16/4 mg); and IM buprenorphine/naloxone (4/1, 8/2, and 16/4 mg). During challenge sessions, physiological status will be recorded continuously and tasks assessing psychomotor, subjective, and objective status will be performed repeatedly.

ELIGIBILITY:
Inclusion Criteria:

* Non-dependent opioid abuser
* Actively abusing opioids by injection

Exclusion Criteria:

* Opioid dependence
* Signs or symptoms of opioid withdrawal, once admitted to residential unit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2000-12; Primary Completion 2002-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Opioid agonist effects | 3.5 hours
Physiologic measures | 3.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States